CLINICAL TRIAL: NCT04161105
Title: Treatment Time-frame Guidelines for Myofascial Dry Needling of Latent Myofascial Trigger Points in the Muscles of the Lower Limb Kinetic Chain.
Brief Title: Treatment Time-frame Guideline for Dry Needling in the Lower Limb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Technology, Carlow (Other)
Responsible Party: Principal Investigator, Darragh O'Meara, Principal Investigator, Institute of Technology, Carlow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DomMSc
Record Dates: First submitted 2019-11-11; First posted 2019-11-13 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Trigger Points
Keywords: Dry needling; Strength; Latent trigger points
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Participants with latent trigger points in rectus femoris (RF) and gluteus maximus (GM) muscles will be stratified evenly into 3 groups (RF dry needling, GM dry needling or control) based on baseline strength. Treatment, data collection and data analysis of all participants will be conducted concurrently.
Who Masked: Outcomes Assessor
Masking Description: The principal investigator will gather data using a force platform and computer software. It will be anonymised and group allocation will be concealed by a second investigator before being individually analysed by the principal investigator. The second investigator will be given the individually analysed data and he/she will sort the individual data into relevant groups for group analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rectus femoris dry needling group (Experimental): The rectus femoris dry needling group will have their strength assessed. They will then receive one treatment of dry needling to a trigger point in their rectus femoris muscle. They will have their strength re-assessed 24, 48 & 72 hours after dry needling.
  Interventions: Procedure: Dry needling
- Gluteus maximus dry needling group (Experimental): The gluteus maximus dry needling group will have their strength assessed. They will then receive one treatment of dry needling to trigger points in their gluteus maximus muscle only. They will have their strength re-assessed 24, 48 & 72 hours after dry needling.
  Interventions: Procedure: Dry needling
- Control (No Intervention): This group will receive no intervention. They will have their strength assessed at baseline and 24, 48 & 72 hour follow-up

INTERVENTIONS:
Procedure: Dry needling — Dry needling is an invasive procedure involving inserting acupuncture needles directly into trigger points within muscles. The needle is partially withdrawn and re-inserted repeatedly to maximally stimulate the muscle and it's fibers.
  Other Names: Myofascial dry needling
  Arms: Gluteus maximus dry needling group; Rectus femoris dry needling group

SUMMARY:
This study evaluates the impact of treating myofascial trigger points with a single session of dry needling on maximal isometric strength in the short term. Two groups will receive dry needling in separate muscle groups and a third group will receive no dry needling.

DETAILED DESCRIPTION:
Dry needling is a effective treatment for myofascial trigger points. It is very common in a sporting environment. Strength is a key aspect of athletic performance. Despite the prevalence of dry needling within a sporting environment, the effects of dry needling on strength remains unknown.

This study will investigate the effects of dry needling on maximal isometric strength with a view to informing clinical practice amongst clinicians working in the elite sport setting.

ELIGIBILITY:
Inclusion Criteria:

* Must have latent trigger points in their rectus femoris and gluteus maximus

Exclusion Criteria:

* Active trigger points in rectus femoris or gluteus maximus
* Participants with current injuries
* History of fibromyalgia or myofascial pain syndrome
* History of blood disorder which prevents dry needling
* Needle phobia
* History of surgery in the last 6 months

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Isometric peak force during the isometric mid-thigh pull | Baseline, 24 hours post intervention, 48 hours post intervention, 72 hours post intervention.
  Measured in newtons. It is the amount of force exerted by pulling against an immovable bar. Peak force is measured as vertical ground reaction by force platforms beneath the participants feet.
Isometric peak rate of force development during the isometric mid-thigh pull | Baseline, 24 hours post intervention, 48 hours post intervention, 72 hours post intervention.
  Measured in newtons per second squared. It is the amount of force exerted by pulling against an immovable bar divided by the amount of time it takes to generate the force. It is measured as vertical ground reaction by force platforms beneath the participants feet.
Relative isometric peak force during the isometric mid-thigh pull | Baseline, 24 hours post intervention, 48 hours post intervention, 72 hours post intervention.
  Measured in newtons per kg body weight. It is the amount of force exerted by pulling against an immovable bar divided by two thirds the participants body weight. Peak force is measured as vertical ground reaction by force platforms beneath the participants feet.
Relative isometric peak rate of force development during the isometric mid-thigh pull | Baseline, 24 hours post intervention, 48 hours post intervention, 72 hours post intervention.
  Measured in newtons per second squared per kg. It is the amount of force exerted by pulling against an immovable bar divided by the amount of time it takes to generate the force divided by two thirds the participants body weight. It is measured as vertical ground reaction by force platforms beneath the participants feet.
Normalised isometric peak rate of force development during the isometric mid-thigh pull | Baseline, 24 hours post intervention, 48 hours post intervention, 72 hours post intervention.
  Measured in newtons per second squared and expressed relative to each participant peak force. It is the amount of force exerted by pulling against an immovable bar divided by the amount of time it takes to generate the force divided by the peak vertical ground reaction force produced during the trial. It is measured as vertical ground reaction by force platforms beneath the participants feet.
Isometric time interval rate of force development during the isometric mid-thigh pull | Baseline, 24 hours post intervention, 48 hours post intervention, 72 hours post intervention.
  Measured in newtons per second squared. It is the amount of force exerted by pulling against an immovable bar divided by the amount of time it takes to generate the force. With values expressed in specific time interval windows (0ms to 50ms, 0-100ms, 0-150ms, 0-200ms, 0-250ms) It is measured as vertical ground reaction by force platforms beneath the participants feet.

CONTACTS AND LOCATIONS:
Overall Officials: Darragh O' Meara, BSc, Principal Investigator — Institute of Technology, Carlow
Locations (1):
- Institute of Technology Carlow, Carlow, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No